CLINICAL TRIAL: NCT02025543
Title: Confounder-Corrected Quantitative Magnetic Resonance Imaging (MRI) Biomarker of Hepatic Iron Content
Brief Title: Confounder-Corrected Quantitative MRI Biomarker of Hepatic Iron Content
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Johns Hopkins University (Other); Stanford University (Other); University of Texas (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2013-1174; A539300 (Other: UW Madison); SMPH/RADIOLOGY/RADIOLOGY* (Other: UW Madison); R01DK100651 (NIH); Protocol Version 12/12/22 (Other: UW Madison)
Record Dates: First submitted 2013-12-12; First posted 2014-01-01 (Estimated); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Iron Overload; Hemochromatosis; Hemosiderosis
Keywords: MRI; Iron overload
MeSH Terms: conditions — Iron Overload; Hemochromatosis; Hemosiderosis | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Patient Group: Subjects with known or suspected iron overload will undergo serum ferritin measurement and an MRI scan.
  Interventions: Device: MRI
- Control Group: Subjects with no known history of iron overload or liver disease will undergo an MRI scan.
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — R2 MRI scan
  Other Names: Magnetic Resonance Imaging

SUMMARY:
The purpose of this multi-site research is to validate a rapid magnetic resonance based confounder-corrected R-2 mapping method as a quantitative imaging biomarker of liver iron concentrations.

DETAILED DESCRIPTION:
This multi-center, multi-vendor study will validate a rapid magnetic resonance-based confounder-corrected R2* mapping method as a quantitative imaging biomarker of liver iron concentration (LIC). Excessive accumulation of iron in various organs, including the liver, which affects both adult and pediatric populations, is toxic and requires treatment aimed at reducing body iron stores. Measurement of LIC is critical for detection and staging of iron overload, and for monitoring iron-reducing chelator therapies that are expensive and have side effects. Magnetic Resonance Imaging (MRI) is a widely available, accessible, and safe technology, and it is very sensitive to the presence of iron in tissue. Translation of an MRI biomarker of liver iron concentration into broad clinical use requires that it is clinically feasible, precise, robust to changes in scan parameters, calibrated to a validated reference standard of LIC, and is reproducible across sites and manufacturers. There are currently no available MRI methods that meet these requirements. R2*-MRI holds the greatest promise to meet these requirements. R2* mapping can be performed very rapidly with whole-liver 3D coverage in a single 20s breath-hold.

Protocol Modification approved to include additional liver susceptibility measurements for approximately 10 participants (already enrolled at the UW) via recently acquired Superconducting Quantum Interference Device (SQUID). The completion of this additional imaging will depend upon the successful set up and installation of this device.

Per a protocol amendment approved on 10/11/21, the investigators are re-opening the study and increasing enrollment for control subjects. Up to 20 control subjects (changed from 5) will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* know or suspected iron overload
* minimum age: Stanford- 8years , University of Wisconsin - 10 years, John Hopkins follow- 10 years, University of Texas-Southwestern - 18 years

Exclusion Criteria:

* contraindication to magnetic resonance imaging

Ages: 8 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants with known or suspected iron overload, plus a control cohort
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2015-08-12 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Calibration curve of liver R2* vs LIC measured by Ferriscan at each of the sites | 1 year
  The hypothesis is that equivalence between R2 measured with different protocols with higher repeatability than standard MRI iron imaging measurement and with linear calibration to liver iron concentration will be demonstrated. This project will be considered a success if the reproducibility of confounder-corrected R2 MRI is established: the hypothesis is that calibrations at all sites will be equivalent.

SECONDARY OUTCOMES:
Precision: Difference in UW-measured R2* vs Average | 2 years
  Repeat scans will be used at each site to determine precision of R2 liver iron concentration. Repeat scans on n=25 subjects per site will be used to determine Bland-Altman 95% limits of agreement (LOA) by plotting the difference in UW-measured R2* vs average.
Diagnostic Accuracy | 2 years
  In addition to correlation with liver iron concentration (technical accuracy), the diagnostic accuracy through receiver operator characteristic curve analysis will also be determined.
Robustness Assessed via Linear Mixed Effects Regression | 2 years
  At each site and field strength, R2* measurements from the eight different protocols will be compared to assess robustness. Robustness will be assessed via linear mixed effects regression.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Reeder, Principal Investigator — University of Wisconsin, Madison
Locations (4):
- United States (4):
  - Stanford University, Palo Alto, California
  - Johns Hopkins University, Baltimore, Maryland
  - University of Texas-Southwestern, Dallas, Texas
  - University of Wisconsin, Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Case report forms will be coded with a unique study identification number and sent to with the coordinating center by courier. Images will be shared shared using secure FTP server.

REFERENCES:
- [Result] Hernando D, Zhao R, Yuan Q, Aliyari Ghasabeh M, Ruschke S, Miao X, Karampinos DC, Mao L, Harris DT, Mattison RJ, Jeng MR, Pedrosa I, Kamel IR, Vasanawala S, Yokoo T, Reeder SB. Multicenter Reproducibility of Liver Iron Quantification with 1.5-T and 3.0-T MRI. Radiology. 2023 Feb;306(2):e213256. doi: 10.1148/radiol.213256. Epub 2022 Oct 4. PMID 36194113